CLINICAL TRIAL: NCT05956431
Title: A Randomized Controlled Clinical Study of Early Application of Levosimendan to Improve Cardiac Dysfunction and Neurological Prognosis in Patients With Cardiac Arrest
Brief Title: RCT Study of Levosimendan Improving Prognosis of Cardiac Arrest
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Du Lanfang, associate professor, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M2023327
Record Dates: First submitted 2023-07-04; First posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Heart Arrest
Keywords: cardiac arrest; Levosimendan Injection; prognosis
MeSH Terms: conditions — Heart Arrest | interventions — Simendan

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levosimendan group (Experimental): The administration scheme of Levosimendan is continuous intravenous infusion at the rate of 0.05-0.2 μg/kg/min for 24 hours, and no load is given to reduce the risk of Hypotension.
  Interventions: Drug: Levosimendan Injection
- Placebo group (Placebo Comparator): The placebo group received continuous intravenous infusion of physiological saline at the rate of 0.05-0.2 μg/kg/min for 24 hours, while also receiving comprehensive cluster therapy with PCAS.
  Interventions: Drug: physiological saline

INTERVENTIONS:
Drug: Levosimendan Injection — The administration scheme of Levosimendan is continuous intravenous infusion at the rate of 0.05-0.2 μg/kg/min for 24 hours, and no load is given to reduce the risk of Hypotension.
  Other Names: Intervention Group
  Arms: Levosimendan group
Drug: physiological saline — The placebo group received continuous intravenous infusion of physiological saline at the rate of 0.05-0.2 μg/kg/min for 24 hours, while also receiving comprehensive cluster therapy with PCAS.
  Other Names: Placebo Group
  Arms: Placebo group

SUMMARY:
This study is intended to use a multicenter, double-blind, superior effect, placebo controlled randomized controlled clinical trial to explore the therapeutic effect of Levosimendan (within 6 hours after the recovery of spontaneous circulation) on mortality and multiple organ dysfunction such as heart and brain in patients with cardiac arrest who have recovered from active Cardiopulmonary resuscitation but have low cardiac output syndrome and coma, and the impact of 30-day mortality and neurological function after cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* 1: Age>18 years old

  2: After active Cardiopulmonary resuscitation, patients with cardiac arrest obtain the recovery of spontaneous circulation (ROSC), which is defined as having palpable arterial pulse lasting for more than 20 minutes

  3: Patients with witnessed cardiac arrest

  4: ROSC lasts for less than 60 minutes

  5: Low cardiac output syndrome after ROSC (LVEF<40%)

  6: Still in a coma after ROSC, Glasgow score<8 points

  7: Complete enrollment within 180 minutes after ROSC

Exclusion Criteria:

* 1: Patients receiving extracorporeal Cardiopulmonary resuscitation

  2: Patients with severe neurological deficits prior to cardiac arrest

  3: Patients with severe renal dysfunction (creatinine clearance rate<30ml/min)

  4: Patients with confirmed or suspected pregnancy

  5: Patients with Intracranial hemorrhage

  6: Patients with end-stage diseases, such as advanced malignant tumors or other severe wasting diseases

  7: Patients who are unwilling to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Cerebral Performance Category (CPC) | On the 30th day after cardiac arrest
  The mortality rate and neurological prognosis at 30 days after cardiac arrest. The evaluation of neurological function adopts CPC score, with CPC 1-2 grading indicating a good prognosis for neurological function and CPC 3-5 grading indicating a poor prognosis for neurological function.

SECONDARY OUTCOMES:
Survival rate | after 1 week of resuscitation
  Survival rate after 1 week of resuscitation was counted
Echocardiography | On the first week after resuscitation
  After enrollment, echocardiography parameters were collected according to the time nodes specified in this research process
Neuron-Specific Enolase (NSE) | On the first week after resuscitation
  After enrollment, NSE was collected according to the specified time points in this study process
Gray-to-White Matter Ratio (GWR) | On the first week after resuscitation
  After enrollment, head CT GWR were collected according to the specified time points in this study process
Serum creatinine | On the first week after resuscitation
  After enrollment, serum creatinine indicators representing renal function were collected according to the specified time

CONTACTS AND LOCATIONS:
Overall Officials: Ma Qingbian, doctor, Study Chair — Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: Yes
The research results will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When the study is fully completed, it can be shared.
Access Criteria: open access